CLINICAL TRIAL: NCT02946697
Title: A Culturally Sensitive Social Support Intervention
Acronym: JLA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: University of California, Los Angeles (Other); Herald Cancer Association (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: PA18-0280; R01CA180896 (NIH); 16402-02 (Other: University of Houston)
Record Dates: First submitted 2016-10-25; First posted 2016-10-27 (Estimated); Last update posted 2024-10-16 (Actual); Status verified 2024-02

CONDITIONS: Breast Cancer; Breast Neoplasms
Keywords: Chinese; cancer survivors; Quality of Life; Social Support
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Enhanced care and wait-list control group (No Intervention): Participants in the control group will receive enhanced usual care while waiting for the JLA program. Participants will be given information booklets in Chinese developed by the American Cancer Society and cover common issues related to breast cancer, various treatments, and life after treatment. Participants will be asked to read through the booklet individually.
- Social support intervention group (Experimental): The intervention is a 7-week program includes educational and peer mentoring support components. The education curriculum provides information on recognizing side effects of treatment and differentiating them from symptoms of cancer recurrence, physical therapy and alternative treatment, stress management, recognizing depression and managing emotional problems, communication with family members, and body image. The peer-support component assigns each participant with a mentor who is a breast cancer survivor. They share their own experience with participants and also make weekly phone calls to mentees during the intervention to provide support and address remaining concerns.
  Interventions: Behavioral: Social support intervention

INTERVENTIONS:
Behavioral: Social support intervention — The social support intervention is a 7-week program includes educational and peer mentoring support components. The education curriculum provides information on recognizing side effects of treatment and differentiating them from symptoms of cancer recurrence, physical therapy and alternative treatment, stress management, recognizing depression and managing emotional problems, communication with family members, and body image. The peer-support component assigns each participant with a mentor who is a breast cancer survivor. They share their own experience with participants and also make weekly phone calls to mentees during the intervention to provide support and address remaining concerns.
  Other Names: JLA
  Arms: Social support intervention group

SUMMARY:
This study is a randomized controlled trial (RCT) to assess the impact of a culturally based social support program (i.e. Joy Luck Academy, JLA) among Chinese American breast cancer survivors.

DETAILED DESCRIPTION:
This study is a randomized controlled trial (RCT) to test the health benefits of an education and peer mentor support intervention. Chinese American breast cancer survivors who have completed primary treatment will be randomly assigned to either the intervention group or a control group to receive enhanced usual care while waiting for the JLA. Health outcomes are assessed at baseline, immediately post intervention, and 1 and 4 months follow-ups.

ELIGIBILITY:
Inclusion criteria:

* self-identified to be comfortable speaking Chinese (Mandarin or Cantonese)
* having a first breast cancer diagnosis of stages 0-III
* having completed primary treatment (surgery, chemotherapy, or radiotherapy) within the last 36 months

Exclusion criteria:

* unable to read or speak Chinese (Mandarin or Cantonese)
* breast cancer diagnosis of stage IV
* live outside of the LA area

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2024-10-14 (Actual); Study Completion 2024-10-14 (Actual)

PRIMARY OUTCOMES:
Change in Quality of life as assessed by Functional Assessment of Cancer Therapy Scale (FACT) | Baseline before intervention and immediately, 1 month, and 4 months after the intervention

SECONDARY OUTCOMES:
Change in depressive symptoms as assessed by CES-D | Baseline before intervention and immediately, 1 month, and 4 months after the intervention
  Depressive symptoms will be measured with the Chinese short-form version (Boey, 1999) of the Center for Epidemiologic Studies Depression Scale (CES-D; Radloff, 1977) as well as two additional items ("I don't want to have contact with people, socialize, or go out at all" and "I have thought about hurting myself") from the Chinese American Depression Scale (CADS-9).
Change in positive affect as assessed by the PANAS | Baseline before intervention and immediately, 1 month, and 4 months after the intervention
Change in fatigue as assessed by FACIT | Baseline before intervention and immediately, 1 month, and 4 months after the intervention
  A short-version (i.e. 6-item) of Functional Assessment of Chronic Illness Therapy-Fatigue scale was used.
Change in stress as assessed by the Perceived stress scale (PSS) | Baseline before intervention and immediately, 1 month, and 4 months after the intervention

OTHER OUTCOMES:
Change in cortisol slope | Baseline before intervention and immediately

CONTACTS AND LOCATIONS:
Overall Officials: Qian Lu, PhD; MD, Principal Investigator — University of Houston
Locations (1):
- Herald Cancer Association, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lu Q, Warmoth K, Chen L, Wu CS, Chu Q, Li Y, Gallagher MW, Stanton AL, Kagawa Singer M, Young L, Loh A. A Culturally Sensitive Social Support Intervention for Chinese American Breast Cancer Survivors (Joy Luck Academy): Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2021 Sep 22;10(9):e30950. doi: 10.2196/30950. PMID 34550088
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org